CLINICAL TRIAL: NCT03069001
Title: Sofosbuvir and Simeprevir Versus Sofosbuvir and Ribavirin in Egyptian Patients With HCV
Brief Title: Sofosbuvir and Simeprevir Versus Sofosbuvir and Ribavirin in Treatment of HCV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sara Abdelhakam, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 958
Record Dates: First submitted 2017-02-23; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: HCV
Keywords: HCV treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sofosbuvir-Simeprevir (Active Comparator): * Sofosbuvir 400 mg orally once-daily.
  * Simeprevir 150 mg orally once-daily.
  * Group A included 50 patients who received sofosbuvir 400 mg orally once-daily plus simeprevir 150 mg orally once-daily for 12 weeks.
  Interventions: Drug: Sofosbuvir-Simeprevir
- Sofosbuvir-Ribavirin (Active Comparator): * Sofosbuvir 400 mg orally once-daily.
  * Ribavirin orally twice-daily (according to body weight: 1000 mg daily in patients with a body weight of <75 kg and 1200 mg daily in patients with a body weight of ≥75 kg).
  * Group B included 40 patients who received sofosbuvir 400 mg orally once-daily plus ribavirin orally twice-daily for 24 weeks.
  Interventions: Drug: Sofosbuvir-Ribavirin

INTERVENTIONS:
Drug: Sofosbuvir-Simeprevir — -Sofosbuvir-Simeprevir group included 50 patients who received sofosbuvir 400 mg orally once-daily plus simeprevir 150 mg orally once-daily for 12 weeks.
  Arms: Sofosbuvir-Simeprevir
Drug: Sofosbuvir-Ribavirin — -Sofosbuvir-Ribavirin group included 40 patients who received sofosbuvir 400 mg orally once-daily plus ribavirin orally twice-daily for 24 weeks.
  Arms: Sofosbuvir-Ribavirin

SUMMARY:
This prospective study was conducted at Ain Shams University Hospital, Internal Medicine, Hepatology and Gastroenterology Department, and Tropical Medicine Department.

To compare the efficacy of the combination of sofosbuvir and simeprevir for 12 weeks with the combination of sofosbuvir and ribavirin for 24 weeks in Egyptian patients with HCV-related Child A cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic HCV infection with a positive HCV RNA level by PCR.

Exclusion Criteria:

* Total bilirubin > 2 mg/dl.
* serum albumin < 2.8 g/dl.
* INR > 1.7.
* platelet count < 50000/mm3.
* serum creatinine > 2.5 mg/dl.
* patients presented by ascites or hepatic encephalopathy.
* patients with evidence of other causes of liver diseases, including hepatitis A, hepatitis B, autoimmune hepatitis, alcoholic liver disease, drug-induced hepatitis, haemochromatosis, Wilson disease or alpha-1 antitrypsin deficiency.
* patients with any advanced systemic disease.
* pregnancy or inability to use effective contraception in females.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Evaluation at end-of-treatment response | 12 weeks
  undetectable HCV-RNA 12 weeks after the completion of therapy by a sensitive HCV-RNA assay